CLINICAL TRIAL: NCT07053280
Title: A Study That Uses an Organized System to Prospectively Collect Uniform Data From a Defined Population
Brief Title: Teleaudiology: Investigating the Online Applicability of Central Auditory Processing Tests
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Azize Arzu KÖROĞLU KOÇYİĞİT, Lecturer, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/61-25; 1919B012103194 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Central Auditory Processing Disorder; Telehealth
Keywords: central auditory processing, dichotic test, Staggered spondee word test, teleaudiology, temporal processing
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Teleaudiological tests — Initially, the FPT, DPT, RGDT, and SSWT were administered face-to-face; one month later, the same tests were repeated via teleaudiology, with the audiologist and participant in separate rooms using identical laptops and headphones, without visual or auditory contact.

SUMMARY:
The aim of this study is to evaluate the feasibility of applying central auditory processing tests online through teleaudiology. In this context, findings will be presented to increase the accessibility of these tests, with the goal of contributing new data to the existing literature on the usability of online tests in clinical practices. Additionally, investigating the applicability of central auditory processing tests on online platforms aims to provide valuable information regarding diagnostic and assessment processes for individuals who face limitations in accessing audiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Air and bone-conduction hearing thresholds better than 20 dB HL were included in the study
* 18-25 years old
* Type A tympanogram
* Mini mental test score : 24-30
* Normal otoscopic examination

Exclusion Criteria:

* Those who did not meet the inclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who underwent face-to-face and teleaudiology central auditory processing tests | November 2021-February 2022
  41 people were included

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For the purpose of confidentiality of the participants, no individual information will be published, only the analysis results will be published.